CLINICAL TRIAL: NCT00657852
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy of Disodium Pamidronate in the Treatment of Bone Loss Associated With Liver Transplant
Brief Title: Efficacy of Pamidronate in the Treatment of Bone Loss Associated With Liver Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Novartis (Industry)
Responsible Party: Dr. Miquel Navasa Anadón, Digestive Diseases Institute, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 99-NV001
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Bone Disease, Metabolic
Keywords: pamidronate,bone loss, liver transplantation
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Pamidronate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pamidronate (Experimental): Single dose of 90 mg disodium pamidronate within days 7-12 and at 3 months after liver transplantation, diluted in 500 ml of 5% glucose serum and administered as a 4-hour continuous intravenous infusion
  Interventions: Drug: Disodium pamidronate
- Placebo (Placebo Comparator): 500 ml of 5% glucoside serum infusions within days 7-12 and at 3 months after liver transplantation and administered as a 4-hour continuous intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Disodium pamidronate — Single dose of 90 mg disodium pamidronate within days 7-12 and at 3 months after liver transplantation, diluted in 500 ml of 5% glucose serum and administered as a 4-hour continuous intravenous infusion
  Other Names: Aredia
  Arms: Pamidronate
Drug: Placebo — 500 ml of 5% glucoside serum infusions within days 7-12 and at 3 months after liver transplantation and administered as a 4-hour continuous intravenous infusion
  Arms: Placebo

SUMMARY:
The aims of this study are to prospectively evaluate the efficacy of two intravenous infusions of pamidronate 90 mg, associated with calcium and calcidiol, in the early post-transplant period, on bone loss in liver transplant recipients, and to asses the safety of this treatment.

DETAILED DESCRIPTION:
Patients diagnosed with chronic advanced liver disease awaiting orthotopic liver transplantation will be eligible to take part in this study.

Patients excluded from the study will be those younger than 18 years, those receiving a multiorgan transplant or retransplant, or patients with a previous allergy to bisphosphonates. Previous treatment with fluoride, estrogens, selective estrogen receptor modulators or bisphosphonates will be another reason for exclusion, as well as therapy with glucocorticoids during the last 6 months before transplantation. None of the patients will have a previous history of disorders, other than liver disease, known to affect bone metabolism.

Study Design and Conduct

The study will be a 1-year prospective, randomized, double-blind, placebo-controlled trial conducted at 10 centers in Spain.

Immunosuppression

All patients will receive microemulsion cyclosporine A (CsA) as primary immunosuppressive agent, in combination with glucocorticoids. Additionally, mycophenolate mofetil will be associated according to the usual clinical practice of each center. In all cases, glucocorticoids will be progressively tapered during the first year.

Intervention

Patients will receive oral calcium (500 mg twice daily) and oral 25-hydroxy vitamin D (16000 UI every 15 days), after informed consent for the study will be obtained and exploratory screening will be done. Within days 7-12 after engraftment, the recruited transplanted patients (will be randomized to either the experimental or placebo group. Patients of the treatment group will receive a single dose of 90 mg disodium pamidronate within days 7-12 and at 3 months after liver transplantation, diluted in 500 ml of 5% glucose serum and administered as a 4-hour continuous intravenous infusion. Patients of the placebo group will receive 500 ml of 5% glucoside serum infusions. Treatment with oral calcium and vitamin D will be maintained for 1 year after transplantation.

Study Endpoints

The primary endpoints of the study will be changes in bone mineral density (BMD), quantified by dual energy X-ray absorptiometry (DXA) and safety of pamidronate by recording adverse events. Secondary endpoints will include the incidence of skeletal fractures, by assessment of radiological vertebral fractures (symptomatic and asymptomatic), and the development of nonvertebral fractures.

Evaluation

Five study visits will be scheduled: before transplantation, within day 7-12 after liver transplantation and at 3, 6 and 12 months after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with chronic advanced liver disease awaiting orthotopic liver transplantation

Exclusion Criteria:

* younger than 18 years
* receiving a multiorgan transplant or retransplant
* previous allergy to bisphosphonates
* Previous treatment with fluoride, estrogens, selective estrogen receptor modulators or bisphosphonates
* therapy with glucocorticoids during the last 6 months before transplantation
* previous history of disorders, other than liver disease, known to affect bone metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2000-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
bone mineral density (BMD), quantified by dual energy X-ray absorptiometry (DXA) | Change during the 1-year of follow up

SECONDARY OUTCOMES:
adverse events | incidence during 1-year of follow-up
incidence of skeletal fractures, by assessment of radiological vertebral fractures (symptomatic and asymptomatic), | 1-year of follow-up
incidence of nonvertebral fractures | 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Navasa, Dr, Principal Investigator — Hospital Clinic i Provincial, Barcelona
Locations (1):
- Hospital Clinic i Provincial of Barcelona, Barcelona, Barcelona, Spain